CLINICAL TRIAL: NCT04426643
Title: Treatment of Urinary Incontinence in Men After Prostatectomy With Autologous Adipose-derived Mesenchymal Stem Cells Mixed With Collagen Gel and Injected Submucousely
Brief Title: Treatment of Urinary Incontinence in Men After Prostatectomy With Autologous Adipose-derived Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: N.N. Alexandrov National Cancer Centre (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSC(UIM)
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence; Prostatectomy
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenchymal stem cells (Experimental): Patients with Urinary incontinence receiving standard treatment plus adipose-derived mesenchymal stem cells
  Interventions: Biological: Autologous adipose-derived mesenchymal stem cells; Other: Standard treatment according to the Clinical protocols
- control (Active Comparator): Patients with Urinary incontinence receiving standard treatment
  Interventions: Other: Standard treatment according to the Clinical protocols

INTERVENTIONS:
Biological: Autologous adipose-derived mesenchymal stem cells — Autologous adipose-derived mesenchymal stem cells mixed with collagen solution injected in submucosal space
  Arms: mesenchymal stem cells
Other: Standard treatment according to the Clinical protocols — Standard treatment according to the Clinical protocols

SUMMARY:
Treatment of patients with urinary incontinence after prostatectomy using injection of autologous adipose-derived mesenchymal stem cells mixed with collagen gel

DETAILED DESCRIPTION:
During the implementation of the project, it is planned to develop a method for the treatment of men urinary incontinence caused by prostatectomy using injection of autologous adipose-derived mesenchymal stem cells mixed with collagen. The positive outlook for the effectiveness of MSCs is due to the following:

* the ability of MSCs to stimulate tissue regeneration
* positive results of preclinical studies of the method of treatment of urinary incontinence in animals.

In study planing to include 5 patients. MSCs will be isolated from adipose tissue, cultured and then transplanted back to the periurethral area by five point injection in rhabdosphincter and submucosal space of urethra using the cystourethroscope. For injection in submucosal space MSCs (20*10^6 cells) will be mixed with collagen solution (3,5% w|w). Follow up patients monitoring will occur at 1，3，6 and 12 months after injection.

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence
* absence of acute inflammatory manifestations in the genitourinary system
* period after prostatectomy is at least 12 months

Exclusion Criteria:

* urethral or bladder malformations
* acute and chronic infectious diseases: HIV, viral hepatitis, tuberculosis
* mental disorders

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of cured patients | 3 months
  Number of patients cured
Number of patients with treatment-related adverse events | 4 weeks
  MSC application related adverse events assessed by blood count, liver and function tests

CONTACTS AND LOCATIONS:
Overall Officials: Igor D Volotovski, Dr, Study Director — Head of the Lab of Institute of Biophysics and Cell Engineering; Sergey A Krasny, Dr, Study Director — Deputy Director for Research of the National Cancer Centre
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No